CLINICAL TRIAL: NCT04997941
Title: Higher Dose taMOxifen in Premenopausal bREast Cancer Patients: a preoperaTive Window Trial (MORE-T Trial)
Brief Title: Higher Dose Preoperative taMOxifen in Premenopausal bREast Cancer Patients
Acronym: MORE-T
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORE-T trial
Record Dates: First submitted 2021-07-23; First posted 2021-08-10 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Premenopausal Breast Cancer; Hormone Receptor-positive Breast Cancer
Keywords: Premenopausal Breast Cancer; Ki-67; Hormone Receptor-positive Breast Cancer; Tamoxifen
MeSH Terms: interventions — Tamoxifen; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen 40mg (Experimental): Tamoxifen 20mg b.i.d - Participants will be treated for 14 days.
  Interventions: Drug: Tamoxifen Oral Product; Diagnostic Test: Assessment of Ki-67; Procedure: Surgery
- Tamoxifen 20mg (Active Comparator): Tamoxifen 10mg b.i.d - Participants will be treated for 14 days.
  Interventions: Drug: Tamoxifen Oral Product; Diagnostic Test: Assessment of Ki-67; Procedure: Surgery

INTERVENTIONS:
Drug: Tamoxifen Oral Product — Experimental arm will have tamoxifen 40mg and active comparator arm will have tamoxifen 20mg for 14 days.
  Other Names: Tamoxifen 40mg vs. 20mg
Diagnostic Test: Assessment of Ki-67 — Paired biopsies (before and after tamoxifen therapy) will be required for the assessment of Ki-67.
Procedure: Surgery — The surgery date should be fixed before randomization. The surgery is to be performed within 1 day after the last dose of study treatment.

SUMMARY:
MORE-T trial is designed to investigate the effect of Tamoxifen 40mg (vs. Tamoxifen 20mg) for 2wks in presurgical setting.

The greater reduction in Ki-67 might be observed in Tamoxifen 40mg arm compared to the Tamoxifen 20mg arm.

Open Label, Phase 2, Randomized with 1:1 allocation

DETAILED DESCRIPTION:
Tamoxifen

* Selective estrogen receptor modulator
* It has been the main endocrine treatment for decades
* Tamoxifen is a major endocrine treatment option, particularly for women who still have a significant ovarian estrogenic activity that cannot be controlled by aromatase inhibitors.
* The prospective clinical trials have shown that tamoxifen 20mg has comparable efficacy against tamoxifen 40mg with fewer toxicities in breast cancer patients. However, most of the trials comparing tamoxifen 20mg and 40mg were done in postmenopausal women.
* Previous studies have suggested that the higher dose of tamoxifen can induce higher serum levels of the drugs, and increasing tamoxifen dose up to 40mg can induce clinical responses in tumors resistant to 20mg of tamoxifen. A recent prospective trial demonstrated that increasing the dose of tamoxifen from 20 mg to 40 mg can compensate for the reduced endoxifen level in intermediate or poor metabolizer tamoxifen metabolizers based on CYP2D6 genotyping.

Ki-67

* Ki-67 antigen, a nuclear antigen, and marker of cell proliferation, is expressed during all cell-cycle phases except for G0, with levels peaking during mitosis.
* Reduction in Ki67 expression is reported to correlate with treatment response to endocrine therapy in ER+ breast cancer, and Ki-67 in short-term neoadjuvant studies has been shown to predict outcome in long-term adjuvant trials.

As the investigators have a higher proportion of young aged, premenopausal breast cancer patients in Korea, the investigators had an opportunity to examine the prognostic impact of young age in breast cancer recurrences and survivals. The institutional database and the Korean nationwide breast cancer registry data have all shown that the poor prognostic effect of a young age was exclusively seen in women with hormone receptor-positive breast cancers, and the effect was potentially due to the resistance to the tamoxifen. As therapeutic options diversify, studies on factors predictive of sensitivity to various endocrine therapies are needed to help select the appropriate treatment for young premenopausal breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically and immunohistochemically confirmed ER+ and HER2- Premenopausal BC patients
2. Tumor size >0.5cm on USG
3. Stage I-IIIA BC and planned curative surgery
4. ECOG 0-2
5. Patients with adequate bone marrow function

   - Hemoglobin > 10 g/dL, Plt > 100,000/mm3
6. Patients with adequate kidney function

   - serum Cr ≤ 1.4 mg/dL
7. Patients with adequate liver function

   * Bilirubin: ≤ 1.5 times of upper normal limit
   * AST/ALT: ≤ 1.5 times of upper normal limit
   * Alkaline phosphatase: ≤ 1.8 times of upper normal limit
8. Patients who decided to voluntarily participate in this trial with written informed consent
9. Premenopausal women : women who has not removed both ovaries, women who had menses in recent 1 year and FSH level is less than 30mIU/ml

Exclusion Criteria:

1. Previous history of ipsilateral invasive breast cancer, in situ lesion
2. Previous history of chemotherapy or endocrine therapy on contralateral BC for the past 2 years
3. Patients who has distant metastasis
4. Patients who is pregnant or breastfeeding
5. Hormon receptor negative BC
6. Her-2 positive BC
7. Diagnosed pituitary adenoma
8. Women who has endometriosis, unknown vaginal bleeding
9. Inability to understand and willingness to sign a written informed consent
10. Patients with endometriosis or unexplained vaginal bleeding
11. Patients with a history of bleeding constitution, coagulopathy, or thromboembolism
12. Patients who have administered a CYP3A inhibitor or inducer, CYP2D6 inhibitor, etc. within 4 weeks prior to randomization

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Ki-67 level | After 14-day of tamoxifen treatment
  Change in Ki67 (percentage of positive tumor cells tested by immunohistochemistry [IHC] - digital Image Analysis ) after a 14-day treatment period compared to baseline.

SECONDARY OUTCOMES:
Changes in Ki67 according to CYP2D6 genotyping | After 14-day of tamoxifen treatment
  Change in Ki67 (percentage of positive tumor cells tested by immunohistochemistry [IHC]) after a 14-day treatment period compared to baseline according to CYP2D6 genotyping.
The proportion of participants with relative decrease from baseline of Ki-67 ≥50% | After 14-day of tamoxifen treatment
  The proportion of participants with relative decrease from baseline of Ki-67 (% positive tumor cells) ≥50%.
AE | After 14-day of tamoxifen treatment
  Adverse events
SAE | After 14-day of tamoxifen treatment
  Serious adverse events
PEPI (Preoperative Endocrine Prognostic Index) score | After 14-day of tamoxifen treatment
  The PEPI score (ranged 0 to 12, lower score mean a better outcome) is the sum of the risk points of the pathological tumor (pT) stage, the pathological node (pN) stage, Ki67 levels and ER status (Allred score).
RFS | 5 years
  Relapse-free survival rate
OS | 5 years
  Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Gon Moon, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea